CLINICAL TRIAL: NCT04195217
Title: " Application of Art Therapy in Oncology: Evaluation of the Symptomatic of Patients Suffering From a Cancerous Disease"
Acronym: ARONCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Perigueux (Other)
Collaborators: University Hospital, Limoges (Other)
Responsible Party: Principal Investigator, Elodie Barbut Paillard, Principal investigator, Centre Hospitalier de Perigueux
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ID-RCB 2018-A03304-51
Record Dates: First submitted 2019-11-08; First posted 2019-12-11 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Therapy-Associated Cancer
Keywords: ONCOLOGY; ART THERAPY
MeSH Terms: conditions — Neoplasms, Second Primary; Neoplasms | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: This is a interventional study at risk and minimal constraints, paramedical, mono-centric, institutional in view of a validation of innovative practices in the care of the patient, excluding health products.
  It is a superiority, randomized, controlled parallel arms study comparing the usual management and usual care associated with art therapy.
Who Masked: Outcomes Assessor
Masking Description: The biostatistician will analyze the two arms blindly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With art therapy (Active Comparator): Art therapy as supportive care in 6 consecutive sessions of cancer treatments with or without additional supportive care
  Interventions: Behavioral: Art therapy
- Without art therapy (No Intervention): 6 consecutive sessions of cancer treatments without art therapy with other supportive care added.

INTERVENTIONS:
Behavioral: Art therapy — When the patient is placed in a treatment room, a nurse or the ARC proposes to complete the questionnaires corresponding to his visit in accordance with the diagram of the investigations, then retrieve the questionnaire and forward it to the art therapist Then, the art therapist intervenes ans propose different Artistic supports : paint, watercolor pencils, pastels, pencils, clay , origami, music in as an accompaniment to artistic creation.
  The workshop runs from 30 minutes to 2:30. It can be cut by doctors and nurses interventions during medical care. The limit of care is set at 2:30 for reasons of concentration of the patient, organization of the service but the patient is an actor of his care, and chooses when the session ends.
  At the end of intervention, the nurse or the ARC proposes at patient to complete the end questionnaire. Theses last are retrieve it and to forward it to the art therapist.
  Arms: With art therapy

SUMMARY:
The purpose of this study is to evaluate the impact of art-therapeutic management on a patient with cancer, during chemotherapy treatment, on the reduction of physical or psychological symptoms.

Art therapy is a non-drug approach that can help some patients cope with the consequences of cancer beyond the care provided.

The common psychosocial difficulties experienced by cancer patients are pain, fatigue, depression, anxiety, drowsiness. In sum, the well-being and quality of life of the patient throughout the illness.

The main objective is to evaluate the impact of art therapy, as a supportive care, on improving the well-being felt after a session of cancer treatments (chemotherapy, immunotherapy, ...), during 6 sessions( around 24 days between 2 sessions) , at patients with a cancer pathology using two questionnaires, one on the evaluation of symptoms (ESAS), the other on the quality of life (FACT-G).

DETAILED DESCRIPTION:
Patients will be randomized into the following groups:

* Group 1: Art therapy as supportive care in 6 consecutive sessions of cancer treatments with or without additional supportive care
* Group 2: 6 consecutive sessions of cancer treatments with or without additional supportive care.

Symptom assessment with the Edmonton Symptom Assessment System (ESAS) is done before and after each treatment session for each patient.

The FACT-G questionnaire on the quality of life at the beginning and the end of the care for the two groups (group benefiting from the art-therapy and group not benefiting from the art-therapy) and a questionnaire on the contribution of art therapy, at the end of care, for the participants of the art-therapy group.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18
* patient cared for on Onco-hematology day with a cancerous pathology
* consent of the patient
* patient affiliated to social Security

Exclusion Criteria:

* patient minor
* patient under legal protection
* patient with too much impairment of vital and / or cognitive functions to participate and understand the study
* patient whose predictable management is less than the follow-up period (6 sessions),
* patient who has already participated in an art therapy session during their lifetime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-03-17 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution well-being felt | Before and after each chimotherapy session - 6 sessions between 6 weeks to 6 months
  The aim is to evaluate the impact of art therapy as a supportive care on the improvement of the well-being felt after a session of cancer treatments (chemotherapy, immunotherapy, ...), during 6 sessions, in patients having a cancerous pathology.
  The primary endpoint is the 6-session average of the difference between the ESAS score associated with the patient's well-being symptom (a symptom of "feeling good" on the ESAS assessment), obtained before and after the treatment session.
  The Edmonton Symptom Assessment System (SESA) is a 9-item symptom rating scale. The quote goes from 0 to 10. A score close to zero means a better result. The comparison of the mean differences between the ESAS score before and after each of the six cancer treatment sessions according to the two randomization groups will be performed using a generalized linear model.

SECONDARY OUTCOMES:
evaluation of all items on the ESAS scale along 6 sessions | Before and after each chemotherapy session - 6 sessions between 6 weeks to 6 months
  Evaluate the impact of art therapy as supportive care on the reduction of ESAS symptoms after one treatment session for 6 sessions.
  Secondary endpoint 1, for each of the other symptoms of the ESAS scale, is pain, fatigue, nausea, depression, anxiety, drowsiness, lack of appetite, difficulty breathing, or other symptoms to be discussed by the patient. , the average over 6 treatment sessions, the difference between the ESAS score associated with the symptom studied, obtained before and after each treatment session.
  The Edmonton Symptom Assessment System (SESA) is a 9-item symptom rating scale. The quote goes from 0 to 10. A score close to zero means a better result. The comparison of the mean differences between the ESAS score before and after each of the six cancer treatment sessions according to the two randomization groups will be performed using a generalized linear model.
evaluation of all items on the ESAS scale between first and last session | 6 sessions between 6 weeks to 6 months
  To determine the impact of the 6 sessions of art therapy as supportive care to cancer treatments on the evolution of symptoms, by the ESAS scale, before the first session of art therapy, and after the last session (6th) The secondary judgment criterion 2 corresponds, for each of the ESAS symptoms, to the difference in ESAS score associated with the symptom studied, before the first and the last treatment session (6th).
  The Edmonton Symptom Assessment System (SESA) is a 9-item symptom rating scale. The quote goes from 0 to 10. A score close to zero means a better result. The comparison of the mean differences between the ESAS score before and after each of the six cancer treatment sessions according to the two randomization groups will be performed using a generalized linear model.
evolution of the Fact G quality of life assessment items | 6 sessions between 6 weeks to 6 months
  To evaluate the impact of the 6 sessions of art-therapy, as supportive care in onco-therapy, on the evolution of the quality of life.
  Secondary endpoint 3 is the difference in total FACT-G quality of life score score between inclusion and the end of the 6 sessions of cancer treatment.
  This questionnaire contains 27 items constructed on a Likert scale with 5 coded response modes: 0 "Not at all" / 1 "A little" / 2 "Moderately" / 3 "A lot" / 4 "Enormously".
  A score is calculated by dimension. These scores range from 0 to 28 where 0 represents a low level of well-being and 28 a high level of well-being. This score corresponds to the sum of the raw scores obtained for each dimension, and varies from 0 (low level) to 108 (good level of general well-being).
art therapy satisfaction questionary | End of 6 session between 6 weeks to 6 months
  Questionnaire (created by the principal investigator) designed to evaluate patient satisfaction, after 6 sessions of art therapy, on this type of therapy as supportive treatment in onco-therapy. It is composed of 5 questions relating to the feeling of art therapy sessions by the patient. They are rated from 0 to 5 (a better score is close to 5) in relation The secondary endpoint 4 is the satisfaction questionnaire for art therapy, performed only in patients in the therapy group by art.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie EP BARBUT PAILLARD, SEARCHER, Principal Investigator — Hospital center of Périgueux
Locations (1):
- Perigueux Hospital Center, Périgueux, Dordogne, France

IPD SHARING:
Plan to Share IPD: No
data sharing characteristics are not yet defined

REFERENCES:
- [Background] Schiltz L, Zimoch A. [Using arts therapies in psycho-oncology: evaluation of an exploratory study implemented in an out-patient setting]. Bull Soc Sci Med Grand Duche Luxemb. 2013;(1):48-71. French. PMID 23808110
- [Background] Gotze H, Geue K, Buttstadt M, Singer S, Schwarz R. [Art therapy for cancer patients in outpatient care. Psychological distress and coping of the participants]. Forsch Komplementmed. 2009 Feb;16(1):28-33. doi: 10.1159/000191211. Epub 2009 Jan 30. German. PMID 19295227
- [Background] Puetz TW, Morley CA, Herring MP. Effects of creative arts therapies on psychological symptoms and quality of life in patients with cancer. JAMA Intern Med. 2013 Jun 10;173(11):960-9. doi: 10.1001/jamainternmed.2013.836. PMID 23699646
- [Background] Nainis N, Paice JA, Ratner J, Wirth JH, Lai J, Shott S. Relieving symptoms in cancer: innovative use of art therapy. J Pain Symptom Manage. 2006 Feb;31(2):162-9. doi: 10.1016/j.jpainsymman.2005.07.006. PMID 16488349
- [Background] Geue K, Goetze H, Buttstaedt M, Kleinert E, Richter D, Singer S. An overview of art therapy interventions for cancer patients and the results of research. Complement Ther Med. 2010 Jun-Aug;18(3-4):160-70. doi: 10.1016/j.ctim.2010.04.001. Epub 2010 May 15. PMID 20688262
- [Background] Bruera E, MacMillan K, Hanson J, MacDonald RN. The Edmonton staging system for cancer pain: preliminary report. Pain. 1989 May;37(2):203-209. doi: 10.1016/0304-3959(89)90131-0. PMID 2748193
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Wood MJ, Molassiotis A, Payne S. What research evidence is there for the use of art therapy in the management of symptoms in adults with cancer? A systematic review. Psychooncology. 2011 Feb;20(2):135-45. doi: 10.1002/pon.1722. PMID 20878827
- [Background] Lefevre C, Ledoux M, Filbet M. Art therapy among palliative cancer patients: Aesthetic dimensions and impacts on symptoms. Palliat Support Care. 2016 Aug;14(4):376-80. doi: 10.1017/S1478951515001017. Epub 2015 Nov 20. PMID 26584521
- [Background] Rhondali W, Lasserre E, Filbet M. Art therapy among palliative care inpatients with advanced cancer. Palliat Med. 2013 Jun;27(6):571-2. doi: 10.1177/0269216312471413. No abstract available. PMID 23685771
- [Background] Conroy T, Mercier M, Bonneterre J, Luporsi E, Lefebvre JL, Lapeyre M, Puyraveau M, Schraub S. French version of FACT-G: validation and comparison with other cancer-specific instruments. Eur J Cancer. 2004 Oct;40(15):2243-52. doi: 10.1016/j.ejca.2004.06.010. PMID 15454249
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- See also: Quality of life of patients with colorectal cancer — http://www.em-consulte.com/en/article/98222